CLINICAL TRIAL: NCT06345001
Title: An Open-label Phase 1 Imaging Study to Evaluate the Biodistribution, Dosimetry, Safety and Pharmacokinetics of BAY 3630942, a 89Zr-labeled Monoclonal Antibody, With a Pre-infusion of BAY 3547922, a Monoclonal Antibody-chelator Conjugate, in Patients With Hepatocellular Carcinoma or Other Select Solid Tumors.
Brief Title: A First-in-Human Study to Learn About How BAY3630942 is Distributed and Processed Inside the Body When Given After BAY3547922 and How Safe it is in People With Liver Cancer or Other Select Solid Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 22261
Record Dates: First submitted 2024-03-28; First posted 2024-04-03 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Hepatocellular Carcinoma (HCC); Solid Tumors
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 - Total mass dose selection (Experimental): Participants with HCC or other select solid tumors will receive a single dose of BAY3630942 after intravenous (IV) administration of a specified dose of BAY3547922. Up to 5 total mass dose levels may be tested.
  Interventions: Drug: BAY3630942; Drug: BAY3547922
- Part 2 - Actinium-225 Dosimetry Estimates (Experimental): Participants with HCC or other select solid tumors will receive the total mass dose level selected in Part 1.
  Interventions: Drug: BAY3630942; Drug: BAY3547922

INTERVENTIONS:
Drug: BAY3630942 — IV, Single administration
Drug: BAY3547922 — IV, Single infusion

SUMMARY:
Researchers are studying a new potential treatment for liver cancer or other select solid cancers.

To do this, researchers have developed a protein, called a monoclonal antibody, which can find and attach itself to another protein present on the surface of cancer cells. This can help the new treatment to specifically target cancer cells.

In this study, researchers want to understand the distribution and processing of this monoclonal antibody in people with liver cancer or other select solid cancers.

Researchers will use the following two forms of monoclonal antibody as study interventions during this study:

* BAY3630942: This is the monoclonal antibody attached to a tracer. A tracer emits radiation that can help researchers track the monoclonal antibody in the body using imaging tests like PET/CT (positron emission tomography / computed tomography). All participants will receive a fixed dose of BAY3630942 during the study.
* BAY3547922: This is the monoclonal antibody without the tracer. Participants may receive different amounts of BAY3547922 during the study.

In this study, participants will not derive therapeutic benefit from receiving BAY3630942 or BAY3547922. However, this study may help researchers develop a new treatment for people with liver cancer or other select solid cancers and find a dose to be tested in future studies.

The main purpose of this first-in-human study is to check how BAY3630942 distributes among different organs in the body and how much of the radiation it emits is absorbed by the organs based on the total dose of BAY3630942 and BAY3547922 given. For this, the researchers will:

* measure the amount of BAY3630942 radiation found in different organs over time.
* measure the amount of BAY3630942 radiation absorbed by different organs.
* use the above information to estimate the amount of radiation that would be absorbed by the same organs from the new potential treatment.

Researchers will also monitor the number and severity of medical problems participants have after receiving BAY3630942 and BAY3547922. These medical problems are also known as "adverse events". Doctors keep track of all medical problems that happen in studies, even if they do not think they might be related to the study interventions.

The study participants will first receive BAY3547922 as an infusion into a vein followed by BAY3630942 as an injection into the same vein. Both interventions will be administered only once, on the same day.

Each participant will be in the study for around 44 days with up to 7 visits to the study clinic which includes:

* a visit up to 14 days before the start of the study to confirm if the participant can take part in the study.
* up to 5 visits during the imaging intervention period. During this period, participants:

  * will receive the study interventions and have blood tests on the first visit,
  * will have imaging and blood tests on the next 3 visits. The tests scheduled for the second visit may be performed during the first visit.
  * may have blood tests on the last visit.
* a follow-up visit to check their health after 30 days of receiving the study interventions.

During the study, the doctors and their study team will:

* check participants' health by performing tests such as blood and urine tests, and check heart health using an electrocardiogram (ECG)
* track and study BAY3630942 using PET/CT imaging tests

As the study interventions are not yet treatments for liver cancer or other select solid cancers, access to BAY3630942 and BAY3547922 after the end of the study will not be required.

ELIGIBILITY:
Inclusion Criteria:

* Participant (male or female) must be 18 years of age inclusive, at the time of signing the informed consent.
* Histologically confirmed HCC or non-invasive diagnosis of HCC according to American Association for the Study of Liver Diseases (AASLD) criteria
* Histologically or cytologically confirmed solid tumors
* Child-Pugh class A and B7
* Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1
* Able to tolerate the study procedures, including 3 PET/CT scans
* Adequate bone marrow, hepatic, and renal function
* Agreed to take proper contraception measures

Exclusion Criteria:

* Impaired cardiac function or clinically significant cardiac disease (i.e., congestive heart failure New York Heart Association [NYHA] Class II, III or IV).
* Patients with arterial thrombotic or embolic events or venous pulmonary embolism within 3 months before the start of study intervention.
* On-going systemic anticancer therapy except continued luteinizing hormone-releasing hormone (LHRH) agonist or antagonists in participants with prostate adenocarcinoma
* Administered a radioisotope within 9 physical half-lives of that radioisotope (24 days for yttrium-90 or 90Y) before administration of the study interventions
* Any local or locoregional therapy of intrahepatic tumor lesions, open biopsy or significant traumatic injury < 4 weeks before administration of the study interventions.
* Known hypersensitivity to human monoclonal antibodies.
* Any condition which, in the opinion of the Investigator, would preclude participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2024-08-26 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Radioactivity concentration (SUVmean, %ID/g) of BAY3630942 in normal organs (including but not limited to kidney, spleen, liver, and bone marrow) as a function of time using 3 post-administration PET/CT scans | Up to 12 days
Zirconium-89 absorbed doses (mGy/MBq) in normal organs | Up to 12 days
Absorbed doses (mGy/MBq) from actinium-225 and daughter radionuclides in critical organs estimated | Up to 12 days
  By using the normal organ biodistribution time-course data of BAY3630942 (with assumptions on actinium-225 daughter radionuclides redistribution to critical organs)

SECONDARY OUTCOMES:
Proportion and severity of adverse events (AEs) after administration of BAY3630942 and BAY3547922 | Up to 30 days
Cmax (from zirconium-89 radioactivity concentration (Bq/g and %ID/kg) as a function of time in blood) | Up to 12 days
  Cmax: Maximum observed concentration
AUC (from zirconium-89 radioactivity concentration (Bq/g and %ID/kg) as a function of time in blood) | Up to 12 days
  AUC: Area under the curve
Cmax (from plasma concentration of total antibody (mg/L and %ID/L) as a function of time) | Up to 12 days
AUC (from plasma concentration of total antibody (mg/L and %ID/L) as a function of time) | Up to 12 days

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - City of Hope - Duarte Cancer Center, Duarte, California
  - University of Southern California (USC) - Norris Comprehensive Cancer Center, Los Angeles, California
  - Biogenix Molecular, LLC, Miami, Florida

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards — https://clinicaltrials.bayer.com/study/22261